CLINICAL TRIAL: NCT03796273
Title: tGLI1 as a Therapeutic Target in Brain Metastases: A Window of Opportunity Study in Breast Cancer Brain Metastases and Primary Gliomas
Brief Title: Ketoconazole Before Surgery in Treating Patients With Recurrent Glioma or Breast Cancer Brain Metastases
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054587; NCI-2018-03087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 91118 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-12-26; First posted 2019-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Astrocytoma; Breast Carcinoma Metastatic in the Brain; Glioma; Invasive Breast Carcinoma; Oligodendroglioma; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Glioma
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma | interventions — Practice Guidelines as Topic; Standard of Care; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ketoconazole) (Experimental): Patients receive ketoconazole PO QD on days 1-4 before standard surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Drug: Ketoconazole
- Arm II (standard surgery) (Active Comparator): Patients undergo standard surgery.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Undergo standard surgery
  Other Names: standard of care; standard therapy
Drug: Ketoconazole — Given PO
  Other Names: Fungarest; Fungoral; Ketoderm; Ketoisdin; Nizoral; Orifungal M; Panfungol; R-41400; Xolegel
  Arms: Arm I (ketoconazole)

SUMMARY:
This trial studies the side effects and how well ketoconazole works before surgery in treating patients with glioma that has come back or breast cancer that has spread to the brain. Ketoconazole is an antifungal drug that may be able to block a protein, tGLI1 and may help to treat brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if ketoconazole alters the tGLI1 activation signature (tGAS) which is consisted of eight validated tGLI1 regulated genes (CD24, CD44, VEGF-A, VEGF-C, VEGFR2, TEM7, OCT-4. and heparanase) in tGLI1 expressing brain biospecimens.

SECONDARY OBJECTIVES:

I. To determine if pre-treatment with ketoconazole, an inhibitor of the tGLI1 pathway in tissue culture and animal models, reduces circulating tGLI1 associated exosomal miRNA expression (miR1290 and miR1246) in brain tumor patients.

II. To describe the safety of ketoconazole when administered peri-operatively to patients with primary and secondary brain tumors.

III. To measure the blood brain penetrance of ketoconazole in serum relative to enhancing brain tissue.

EXPLORATORY OBJECTIVES:

I. To measure blood brain penetration of ketoconazole in serum relative to cerebrospinal fluid (CSF) and serum relative to non-enhancing brain tissue (exploratory recurrent glioma patients only).

II. To compare tGLI1 expression and pathway modulation with ketoconazole pre-treatment in patients with recurrent gliomas relative to breast cancer brain metastases (BCBM).

III. To determine the overall survival and toxicity outcomes for patients that continue ketoconazole after surgery, at the discretion of the treating physician.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ketoconazole orally (PO) once daily (QD) on days 1-4 before standard surgery in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo standard surgery.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a history of:

  * Histologically confirmed primary breast cancer including primary invasive and metastatic breast cancers with imaging findings consistent with brain metastasis. In the event that a patient presents with an initial diagnosis of metastatic breast cancer with imaging findings of a new brain metastases and unequivocal imaging findings of a primary breast cancer, consideration for study enrollment requires approval from the study chair (primary cohort)

OR

* Histologically confirmed primary glioma including astrocytoma or oligodendroglioma of any World Health Organization grade with imaging findings consistent with recurrent or progressive disease (exploratory cohort). Patients with ependymoma will not be included.

  * Subjects must be undergoing surgical resection for clinical purposes with anticipated resection of at least 300 mg of tissue.
  * Patients with any prior number of radiation (including brain radiation), chemotherapy, or surgical interventions will be eligible for this protocol.
  * The effects of ketoconazole on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Subjects with contraindication to ketoconazole including:

  * Prior allergic reaction or intolerance of ketoconazole
  * Known active hepatitis
  * QTc prolongation (based on electrocardiography [EKG] obtained within 21 days of enrollment, with a threshold of >450 ms in males and >470 ms in female)
  * Known liver cirrhosis will be excluded from enrollment
  * Positive serum pregnancy test within 21 days of enrollment
* Subjects currently taking medications that are included in the contraindicated concurrent medications section of the Food and Drug Administration (FDA) approved indications for ketoconazole will be required to complete a seven day wash out period prior to consideration for enrollment.
* Subjects for whom collection of blood, or tissue samples is unsafe or clinically inadvisable.
* Pregnant women are excluded from this study because ketoconazole is a Class B agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ketoconazole, breastfeeding should be discontinued if the mother is treated with ketoconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
tGLI1 activation signature 8 (t-GAS 8) | Up to 30 days after surgery
  The primary outcome of this study is modulation of the tGLI1 pathway as assessed by the tGLI1 activation signature 8 (t-GAS 8) [29, 40]. t-GAS 8 consists of eight validated tGLI1 regulated genes (CD24, CD44, VEGF-A, VEGF-C, VEGFR2, TEM7, OCT-4. and heparanase) and is measured using qPCR in patients whose brain tissue expresses tGLI1 (by IHC). The distribution of the tGAS will be examined and transformed to approximate the conditional normality assumption if necessary. Analysis of variance (ANOVA) methods will be used to determine the effects of different factors of interest (e.g., treatment or tumor type) on the outcomes measured.

SECONDARY OUTCOMES:
tGLI1 pathway activation | Up to 30 days after surgery
  tGLI1 pathway activation will be compared between treatment groups using ANOVA as described for the analysis of primary objective.
Incidence of adverse events (AEs) | Up to 30 days after surgery
  The safety of ketoconazole will be defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 criteria and determined by adverse event proportions. The adverse event proportions will be compared between treatment groups using chi-squared tests. If feasible, a logistic regression model will be used to detect whether the adverse event proportion is higher in the treatment group after adjusting for the tumor type.
Blood brain penetrance of ketoconazole in serum relative to enhancing brain tissue | Up to 30 days after surgery
  The analysis will be the same as that for the analysis of primary objective.

OTHER OUTCOMES:
Serum ketoconazole concentrations in Cerebrospinal Fluid (CSF) | Up to 30 days after surgery
  Measured using mass spectroscopy. The analysis will be the same as that for the analysis of primary objective. If the sample size is too small, the nonparametric approach will be considered as the primary analysis.
Serum ketoconazole concentrations in enhancing brain tissue | Up to 30 days after surgery
  Measured using mass spectroscopy. The analysis will be the same as that for the analysis of primary objective. If the sample size is too small, the nonparametric approach will be considered as the primary analysis.
Serum ketoconzcole concentrations in unenhancing brain tissue | Up to 30 days after surgery
  Measured using mass spectroscopy. The analysis will be the same as that for the analysis of primary objective. If the sample size is too small, the nonparametric approach will be considered as the primary analysis.
Changes in tGLI1 signaling pathway | Baseline up to 30 days after surgery
  Will be calculated and compared between treatment groups. Ideally analysis of covariance should be done. However, due to the small sample size, ANOVA as described for the primary analysis approach or the 2-sample t test will be used. If needed, non-parametric approaches will be used instead.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03796273/ICF_000.pdf